CLINICAL TRIAL: NCT07280611
Title: The Hering-Breuer Reflex in Bilateral Lung Transplant Patients
Acronym: HB-DLTX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Giacomo Grasselli, Head of department of Anestesia and Intensive care unit, Policlinico Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ID 5483
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Hering-Breuer Reflex
Keywords: Hering-Breuer reflex; Bilateral Lung Transplant

STUDY DESIGN:
Intervention Model Description: The study will be conducted on two groups of subjects:
  * Patients admitted to the Intensive Care Unit for post-operative care following bilateral lung transplantation (Group 1);
  * Patients admitted to the Intensive Care Unit for post-operative care or monitoring after non-thoracic surgery (Group 2 - control group)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral Lung Transplant patients (Experimental): This group include patients admitted to the Intensive Care Unit for post-operative care following bilateral lung transplantation during the weaning phase from mechanical ventilation. The following patients will be excluded: minors, those undergoing retransplantation, single-lung transplantation or urgent lung transplantation; patients with respiratory system compliance < 30 mL/cmH2O; haemodynamically unstable patients and those at increased risk of bleeding due to nasogastric tube placement.
  Interventions: Device: Nasogastric tube placement and elicitation of Hering-Breuer reflex
- Non-thoracic surgery patients (Active Comparator): This group include patients admitted to the Intensive Care Unit for post-operative care or monitoring after non-thoracic surgery. The following patients will be excluded: minors, those who had undergone previous lung transplant or thoracic surgery; patients with respiratory system compliance < 30 mL/cmH2O; haemodynamically unstable patients; those at increased risk of bleeding due to nasogastric tube placement and patients with contraindications to nasogastric tube placement.
  Interventions: Device: Nasogastric tube placement and elicitation of Hering-Breuer reflex

INTERVENTIONS:
Device: Nasogastric tube placement and elicitation of Hering-Breuer reflex — Enrolled patients will have a nasogastric tube placed, through which diaphragmatic electrical activity will be measured. Patients will be ventilated in pressure support mode with an expansion breath delivered at a maximum pressure of approximately 30 cmH2O in order to elicit the Hering-Breuer Reflex. Diaphragmatic electrical activity, timing, volumes and pressures will then be analyzed before and after the expansion breath over a 10 minute period, testing two levels of PEEP (8 and 12 cmH2O).

SUMMARY:
The goal of this clinical trial (non-pharmacologic, single-center) is to determine whether the Hering-Breuer inflation reflex is preserved-and how it is modulated by end-expiratory pressure-in adult intensive-care patients who have undergone bilateral lung transplantation.

The study will enroll men and women ≥ 18 years admitted to the ICU during the early weaning phase and will include a comparison group of intubated ICU patients after major non-thoracic surgery.

The main questions it aims to answer are:

* Is the Hering-Breuer reflex (measured as the ratio THBR/TSPONT) absent or attenuated in double-lung-transplant recipients?
* Does changing the level of positive end-expiratory pressure (PEEP 8 vs 12 cmH₂O) influence the reflex?

Comparison group: Researchers will compare the transplant arm (post-bilateral lung transplantation) with the control arm (post-operative, non-thoracic surgery patients) to see whether loss or blunting of the reflex-and its response to PEEP-differs between the two cohorts.

Participants will:

* Have a nasogastric catheter with embedded electrodes positioned to record the electrical activity of the diaphragm (EAdi).
* Be ventilated in pressure-support mode at two preset PEEP levels (8 cmH₂O and 12 cmH₂O) during the weaning phase.
* Receive one standardized high-volume insufflation at ~30 cmH₂O in each PEEP condition to elicit the reflex, while EAdi, airway pressures, inspiratory/expiratory times, and tidal volumes are recorded for 10 minutes per level.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years;
* Both sexes;
* For group 1: patients admitted to the Intensive Care Unit after undergoing bilateral lung transplantation, during respiratory weaning;
* For group 2: patients admitted to the Intensive Care Unit for support or monitoring after non-thoracic surgery, who will arrive intubated.

Exclusion Criteria:

For group 1, patients meeting at least one of the following criteria will be excluded:

* Re-transplantation or single-lung transplantation;
* Urgent lung transplantation;
* Post-transplant respiratory system compliance < 30 mL/cmH₂O;
* Hemodynamic instability (defined as the presence of one or more of the following: plasma lactate > 4 mmol/L, need for vasoactive support with norepinephrine and/or epinephrine at a dose > 0.05 mcg/kg/min, systolic arterial pressure < 80 mmHg);
* Increased risk of bleeding related to the placement of a nasogastric tube due to coagulopathy or severe thrombocytopenia (INR > 2 and platelets < 70,000);
* Pregnancy

For group 2, patients presenting with one or more of the following criteria will be excluded:

* Postoperative respiratory system compliance < 30 mL/cmH₂O;
* Hemodynamic instability (defined as the presence of one or more of the following: plasma lactate > 4 mmol/L, need for vasoactive support with norepinephrine and/or epinephrine at a dose > 0.05 mcg/kg/min, systolic arterial pressure < 80 mmHg);
* Contraindications to nasogastric tube placement (gastroesophageal surgery within the last 3 months, gastroesophageal bleeding in the previous 30 days, esophageal varices, facial trauma);
* Increased risk of bleeding related to the placement of a nasogastric tube due to coagulopathy or severe thrombocytopenia (INR > 2 and platelets < 70,000);
* History of lung transplantation or major thoracic surgery;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
THBR/TSPONT ratio | At the enrollment
  Comparison of the ratio between the diaphragm electrical activation time after a high-volume breath aimed at eliciting the HBR (THBR) and a spontaneous breath (TSPONT), i.e., the THBR/TSPONT ratio, between patients who underwent bilateral lung transplantation and those who underwent non-thoracic surgery.

SECONDARY OUTCOMES:
The variation of the THBR/TSPONT ratio as a function of PEEP | At the enrollment
  Variation of the THBR/TSPONT ratio calculated at two different PEEP levels (8 and 12 cmH₂O) in patients who underwent bilateral lung transplantation and in those who underwent non-thoracic surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Michigan, Italy

IPD SHARING:
Plan to Share IPD: Yes